CLINICAL TRIAL: NCT03199937
Title: Behavioral and Neural Outcomes of a New Executive Function Treatment for Transition-age Youth With ASD
Brief Title: Executive Function Intervention for High School Students With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Principal Investigator, Cara Pugliese, Principal Investigator, Children's National Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23MH110612-01 (NIH); OAR Innovative Research Award (Other: Organization for Autism Research)
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Executive Functioning; Intervention; Flexible; Unstuck; Transition; Behavior; High school; Problem Solving; Self-Control; Coping
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior; Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor and observers will be blind to the treatment. Classroom observations will be conducted by "partially blind classroom observers." Though the observer will not be told which schools are assigned to which treatment condition, we found that in our last trial occasionally an observer saw treatment materials that suggested which treatment the school had been assigned to. We will make every effort to minimize this, but it may occasionally happen. The pre-post direct child assessments will also be conducted by treatment-blind assessors, as much as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Futures (Experimental): Flexible Futures uses cognitive behavioral therapy (CBT) techniques to target flexibility and planning by teaching core skills through personal goals chosen by students during treatment. Flexible Futures focuses on key functions needed for college success, such as: intrinsic motivation, how to implement skills socially, how thoughts and feelings affect planning and flexibility, self-advocacy skills necessary to promote independence, application of flexibility and organization scripts and strategies in the service of a long-term goal, and management of time and priorities. Guided practice begins with concrete interventionist support, and moves to interventionist cueing, self-cueing, and finally automatic use of the skills without support. Generalization is maximized with school staff as interventionists, parent training, home and classroom extension activities, and role-playing use of strategies in novel situations. Motivation is developed using student choice and natural motivators.
  Interventions: Behavioral: Flexible Futures
- Waitlist control group (Active Comparator): Current standard of care
  Interventions: Other: Current standard of care

INTERVENTIONS:
Behavioral: Flexible Futures — Flexible Futures is a novel and innovative cognitive-behavioral treatment that directly addresses executive function and self-regulation deficits in ASD. Flexible futures targets flexibility and planning through self-regulatory scripts that are consistently modeled and reinforced. Scripts compensate for the inner speech and organization/integration deficits in ASD, and are practiced repeatedly to achieve automaticity. Content focuses on key functions needed for college success, such as: intrinsic motivation, how to implement skills socially, self-advocacy skills application of flexibility and organization scripts and strategies in the service of a long-term goal, and management of time and priorities.
  Arms: Flexible Futures
Other: Current standard of care — Flexible Futures will be compared to a social skills treatment as usual that capitalizes on current standard of care provided by local school districts.
  Arms: Waitlist control group

SUMMARY:
The purpose of this project is to test the effectiveness of a novel school-based intervention targeting executive function skills, including flexibility and planning, in college-track, transition-age youth with ASD. Evaluating treatment change through behavior and brain activity provides important information on how the treatment works and who will best benefit from it.

DETAILED DESCRIPTION:
With half of the $3.2 million lifetime per capita cost of autism spectrum disorder (ASD) attributable to care and productivity loss during adult life, the Interagency Autism Coordinating Committee has identified a pressing need to improve adult outcomes. Even in individuals without intellectual disability who make up 2/3 of children with ASD, as few as 9% reach full functional independence as adults. Failure in college is related to weaknesses in executive function (EF), specifically with flexibility and planning. As such, the transition from high school is a period of amplified risk characterized by poor educational and vocational attainment that persists in adulthood. EF problems are pivotal targets for intervention because they are common, linked to independence, and responsive to treatment in younger children. There are three barriers to treatment outcome research in transition-aged youth with ASD: (1) a lack of proven EF treatments for this age, (2) pervasive failure to generalize skills learned in the clinic to real-world settings, and (3) inadequate objective measures of outcome. This proposal tests the effectiveness of Flexible Futures a new phenotype specific, cognitive behavioral EF intervention to increase flexibility and planning skills for college-track high school students with ASD. It is novel and innovative because its use of translational methods comprehensively evaluates treatment change at the behavioral, cognitive, and neural level.

Cognitive flexibility and planning are impaired in ASD, linked to core ASD symptoms, and embedded in anomalies of brain structure and function. Individuals with ASD fail to activate local cortical regions such as dorsolateral prefrontal cortex (DLPFC) and anterior cingulate cortex (ACC) on set-shifting (flexibility) tasks and show global abnormalities in the default mode, salience, and attentional networks associated with EF problems in attending to important information and implementing goal-directed behavior. In typical development, greater segregation between and greater connectivity within these networks is associated with better cognitive and behavioral regulation. Dr. Pugliese aims to determine whether treatment change can be objectively measured in the brain using functional MRI (fMRI). This cutting edge methodology is critical to identifying processes of treatment change at the neural level, consistent with the NIMH Research Domain Criteria framework, and may yield findings that impact the large variety of psychiatric and developmental disorders linked to EF deficits. Specifically, this study aligns with NIMH K23 guidance soliciting proposals for the development of pilot studies of novel treatments eliciting mechanisms of change.

AIM 1: Refine the Flexible Futures treatment manual and test acceptability, feasibility, and effectiveness in a school setting.

Dr. Pugliese will refine the Flexible Futures manual based on expert opinion and feedback from our in-clinic pilot via an iterative process and run a school-based trial comparing Flexible Futures to social skills treatment. It is hypothesized that intervention acceptability, feasibility, and fidelity will reach an 80% benchmark (H1.1) and students who receive Flexible Futures will show improved EF flexibility and planning abilities in laboratory, school, and home settings post-treatment and at 5-month follow up compared to students who receive treatment as usual (H1.2).

AIM 2: Identify neural correlates of treatment change using fMRI.

Task-evoked and resting-state activation of prefrontal cortex networks will be assessed pre-/post-intervention. It is hypothesized that post-treatment, students receiving Flexible Futures will display increased (normalized) DLPFC and ACC activation during a well-established set-shifting task compared to those receiving social skills training (H2.1), and that activation will be positively correlated with behavioral/cognitive measures of EF (H2.2). It is also hypothesized that post-treatment, students receiving Flexible Futures will display increased connectivity within, and decreased connectivity across default mode, salience, and attentional networks compared to the control group (H2.3).

AIM 3: Identify biomarkers of later EF outcomes at the behavioral, cognitive, and neural level.

Baseline data will be combined across participants to provide a comprehensive EF profile in transition-age youth and identify predictors of later EF and global outcomes. It is hypothesized that baseline measures of EF (behavioral/ cognitive); DLPFC/ACC activation; and greater connectivity within and greater segregation between salience, attentional and default mode networks (neural) will all predict EF outcome and adaptive function. (H3.1).

Significance: Establishing the first effective school-based EF treatment for high-schoolers will provide critical and generalizable transition-related support, and a model for treatment in other prevalent disorders with known EF deficits (e.g. ADHD, anxiety). This training award will launch me toward Dr. Pugliese's ultimate career goals of 1) developing and implementing innovative interventions personalized for specific cognitive profiles, 2) developing school-based treatments to overcome disparities in access to healthcare; and 3) utilizing treatment studies as vehicles to identify biomarkers and provide insight into neural correlates of treatment change.

ELIGIBILITY:
Inclusion Criteria:

* College-track high school students
* Ages 14-22
* Verbal IQ estimate of ≥ 90 on the Wechsler Abbreviated Intelligence Scale-2
* Clinical diagnosis of ASD OR school classification of autism confirmed by clinical impressions and the Social Responsiveness Scale-Revised total score ≥ 65. If the research staff feels that clinical impressions indicate a diagnosis, but parent report is below threshold, the Autism Diagnostic Observation Schedule-2 will be completed.

Exclusion Criteria:

* Bipolar disorder, schizophrenia, or major depression that is currently preventing from participation in classroom activities
* MRI exclusion: contraindication (metal implant or medical device) for MRI

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2015-07-11 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Behavior Rating Inventory of Executive Function (BRIEF)- Self-Report Form (Gioia, Isquith, Guy & Kenworthy, 2000). | On average, 8 and 13 months
  This self-report measure has 55 items with seven clinical scales and three validity scales. It is normed for adolescents between 11 and 18 years of age. Items were developed to capture everyday behaviors associated with EF and tap seven domains: Inhibit, Self-Monitor, shift, Emotional Control, Task Completion, Working Memory, and Plan/Organize. The BRIEF is standardized with normative data expressed as T scores (mean=50; SD=10). Internal consistency is high, with index coefficients in the mid .90s to high .90s, while test-retest stability coefficients for the clinical scales ranged from .67-.79 within the standardization subsample. The individual scales and summary indexes were correlated in various clinical samples with other measures of attentional and behavioral functioning (Behavior Assessment Scales for Children, Child Behavior Checklist, ADHD-RS-IV, Conners 3), providing evidence of convergent and divergent validity.
  Safety Issue: No
Change in Challenge Task (CT) scores | On average, 8 and 13 months
  The Challenge Task is an unpublished, un-normed measure designed by the study staff to measure flexibility and planning in a social context with standardized tasks (Anthony & Kenworthy, 2012). It is a 20-minute play interview that challenges children to be flexible and planful in the context of three activities with an examiner. Specific challenges are posed, and the child's flexibility and planning are scored on a 3-point scale for each task. The scale has task-specific behavioral markers to guide. The CT yields average Flexibility and Planning scores (higher scores indicate greater impairment). Reliability observations will be completed with a second coder for 25% of the videotapes. Examiners in a previous trial achieved interrater agreement >90%, and we will maintain that same standard for the current project.
  Safety Issue: No
Change in Wechsler Abbreviated Scale of Intelligence- Second Edition (WASI-II, Wechsler, 2011), block design subtest | On average, 8 and 13 months
  The WASI-II is an estimate of intelligence, comprised of four subtests, which takes 30-45 minutes to administer. It is a well-standardized task with normative data for ages 6-90. Subtests include the Block Design subtest, the Similarities subtest, the Matrix Reasoning subtest, and the Vocabulary subtest. Performance on each subtest is represented as a T score (mean=50; SD=10), with higher scores indicating better performance. Overall IQ is calculated from a composite of all four subtests and is represented as a standard score (mean=100; SD=15). The entire WASI-2 will be completed at the Baseline Evaluation to identify full-scale IQ and verbal age (based on the vocabulary subtest). Subsequently, the Block Design subtest only will be completed at the Post-Treatment and Long-term Follow-up Evaluations.
  Safety Issue: No
Change in Delis-Kaplan Executive Functioning System (DKEFS; Delis, Kaplan, and Kramer, 2001), Sorting subtest | On average, 8 and 13 months
  The DKEFS is a standardized measure of executive functioning skills and in normed for ages eight through adulthood. The Sorting Subtest particularly measures flexibility. The DKEFS will be completed both at the Baseline and, the Post-Intervention Evaluation as measure of outcome. It takes approximately 10 minutes to administer, and although specific data were not available, the measure has been well documented across several neuropsychological studies to have evidence of reliability and validity.
  Safety Issue: No
Change in Tower of London-Drexel (TOL-DX; Culbertson & Zillmer, 2000) scores | On average, 8 and 13 months
  TOL-DX measures multiple EFs such as planning, inhibition, and working memory. It requires the subject to work step-by-step to copy a pattern of beads on pegs using the least number of moves possible. The total-moves score will be measured as an omnibus measure of EF. Results are reported as standard scores (M = 100; SD = 15).
  Safety Issue: No
Change in Adaptive Behavior Assessment System-Second Edition (ABAS-2) | On average, 8 and 13 months
  (ABAS-II; Harrison and Oakland 2003) is a measure of adaptive behavior with national standardization samples representative of the English speaking US population. The informant report adult form of the ABAS-2(Harrison and Oakland 2003) used in the present study was standardized on an age stratified sample and provided information in the areas of Conceptual (including Communication, Functional Academics, Self-Direction), Social (including not only Social but also Leisure), and Practical (including Community Use, Home Living, Health and Safety, Self-Care) Skills, all of which are presented as norm-referenced standard scores (M = 100; SD = 15) and were used as correlates of interest in the present study.
  Safety Issue: No
Social Responsiveness Scale-Second Edition (SRS-2; Constantino and Gruber 2012) | On average, 8 and 13 months
  The SRS-2 is a 65-item informant report of autistic traits rated on a 4-point Likert Scale (0-3 points). Higher scores indicate more autistic traits; T-scores ≥ 65 (i.e., 1.5 SDs ≥ the population mean of 50) suggest clinically significant autistic traits. The SRS-2 scoring is aligned with DSM-5 criteria for diagnosis of an ASD. The update includes the creation of two higher order indices that correspond to the two symptom domains of ASD: Social Communication and Interaction (SCI) and Restricted Interests and Repetitive Behavior (RRB). Informants provided a single SRS-2 rating for each child in this study. The SRS-2 will be completed at Baseline and Post-Intervention testing.
  Safety Issue: No
Change in Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2)- Parent Form (Gioia, Isquith, Guy & Kenworthy, 2015). | On average, 8 and 13 months
  This parent-report measure contains 63 items with nine clinical scales and three validity scales. It is normed for children ages 5-18. Items were developed to capture everyday behaviors associated with EF and tap nine domains including: Inhibit, Self-Monitor, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Task-Monitor, and Organization of Materials. It is a standardized questionnaire with normative data and standardized scores expressed as T scores (mean=50; SD=10). Internal consistency is high, with index coefficients above .90, while test-retest stability coefficients for the clinical scales ranged from .67-.92 within the parent standardization subsample. The individual scales and summary indexes of the BRIEF-2 were correlated in various clinical samples with other measures of attentional and behavioral functioning (BASC, CBCL, ADHD-RS-IV, Conners 3), which collectively provided evidence of convergent and divergent validity. Safety Issue: No
Flexibility and Planning Interference Scale | On average, 8 and 13 months
  To meet the needs of the current study by addressing the issue of flexibility more specifically, we will modify the BRIEF to include 14 additional unpublished, unnormed "Flexibility" and "Interference" items. These items will assess how much flexibility impacts the child's and family's life. The items will use a 0-3 scale (0-No Interference, 1-Mildly interfering , 2-Moderately Interfering, 3- Severely Interfering) and will ask about behavior observed during the past two weeks (example: "How much do difficulties with flexibility interfere with or disrupt everyday activities (self-care, school, etc.?)") Safety Issue: No
The Swanson, Kotkin, Agler, M-Flynn, and Pelham Scale (SKAMP, Swanson, 1992) | On average, 8 and 13 months
  The SKAMP is a teacher rating scale that takes 5 minutes to complete and assesses impairment from classroom behaviors associated with executive function in adolescents. Although our study uses a modified form of the SKAMP for which reliability and validity data are unavailable, previous community-based trials of the SKAMP showed evidence of high internal consistency, with reliabilities of .98 for overall SKAMP scores, .96 for Deportment (Behavior), and .95 for Attention. The SKAMP was found to be strongly correlated to both parent and teacher versions of the Swanson, Nolan, and Pelham-IV (SNAP-IV; r = .93 and .79 for Inattention and Hyperactivity/Impulsivity). Teachers rate the severity of 10 common behaviors on a 4-point scale, including 6 items related to attention and 4 items related to problematic behavior.
  Safety Issue: No
Classroom Observations | On average, 8 and 13 months
  To further assess functional improvement, at least two 15-minute classroom observations will be conducted by an intervention-blind research assistant (who has achieved reliability on coding criteria) for every study participant. They will occur randomly during the academic school day, but not during Flexible Futures small group sessions or Social Skills training. The following behaviors will be coded for children in this study: Reciprocity, Following Rules, Transitions, Gets Stuck, Negativity/Overwhelm, and Classroom Participation. During the classroom observations, the following behaviors will be coded for the teacher's behavior: Flexibility, Planning/Organizing, Provides Clear Instructions/ Expectations, Actively Uses Visual Support, References Classroom Rules, Maintains Positive Praise: Command/Correction ratio and Uses Reward System.
  Safety Issue: No
Cognitive Flexibility Task | On average, 8 and 13 months
  A task-based fMRI procedure will be used to detect pre-to-post treatment change. Participants will classify pairs of stimuli (objects and pictures) on the basis of how well they "go together" and respond with an appropriate button press. The specific task may change based on pilot results but will be similar to what is proposed.
  Safety Issue: No

CONTACTS AND LOCATIONS:
Overall Officials: Cara E Pugliese, Ph.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pugliese CE, White SW. Brief report: problem solving therapy in college students with autism spectrum disorders: feasibility and preliminary efficacy. J Autism Dev Disord. 2014 Mar;44(3):719-29. doi: 10.1007/s10803-013-1914-8. PMID 23963592
- [Background] Pennington BF, Ozonoff S. Executive functions and developmental psychopathology. J Child Psychol Psychiatry. 1996 Jan;37(1):51-87. doi: 10.1111/j.1469-7610.1996.tb01380.x. PMID 8655658
- [Background] Frith U. Why we need cognitive explanations of autism. Q J Exp Psychol (Hove). 2012;65(11):2073-92. doi: 10.1080/17470218.2012.697178. Epub 2012 Aug 21. PMID 22906000
- [Background] Ganz ML. The lifetime distribution of the incremental societal costs of autism. Arch Pediatr Adolesc Med. 2007 Apr;161(4):343-9. doi: 10.1001/archpedi.161.4.343. PMID 17404130
- [Background] Interagency Autism Coordinating Committee. The 2011 Interagency Autism Coordinating Committee Strategic Plan for Autism Spectrum Disorder Research.; 2011.
- [Background] Farley MA, McMahon WM, Fombonne E, Jenson WR, Miller J, Gardner M, Block H, Pingree CB, Ritvo ER, Ritvo RA, Coon H. Twenty-year outcome for individuals with autism and average or near-average cognitive abilities. Autism Res. 2009 Apr;2(2):109-18. doi: 10.1002/aur.69. PMID 19455645
- [Background] Gobbo K, Shmulsky S. Faculty Experience With College Students With Autism Spectrum Disorders: A Qualitative Study of Challenges and Solutions. Focus Autism Other Dev Disabl. 2013;29(1):13-22. doi:10.1177/1088357613504989.
- [Background] Taylor JL, Mailick MR. A longitudinal examination of 10-year change in vocational and educational activities for adults with autism spectrum disorders. Dev Psychol. 2014 Mar;50(3):699-708. doi: 10.1037/a0034297. Epub 2013 Sep 2. PMID 24001150
- [Background] Hume K, Loftin R, Lantz J. Increasing independence in autism spectrum disorders: a review of three focused interventions. J Autism Dev Disord. 2009 Sep;39(9):1329-38. doi: 10.1007/s10803-009-0751-2. Epub 2009 May 9. PMID 19430897
- [Background] Hill EL. Executive dysfunction in autism. Trends Cogn Sci. 2004 Jan;8(1):26-32. doi: 10.1016/j.tics.2003.11.003. PMID 14697400
- [Background] Pugliese CE, Anthony L, Strang JF, Dudley K, Wallace GL, Kenworthy L. Increasing adaptive behavior skill deficits from childhood to adolescence in autism spectrum disorder: role of executive function. J Autism Dev Disord. 2015 Jun;45(6):1579-87. doi: 10.1007/s10803-014-2309-1. PMID 25398602
- [Background] Kenworthy L, Anthony LG, Naiman DQ, Cannon L, Wills MC, Luong-Tran C, Werner MA, Alexander KC, Strang J, Bal E, Sokoloff JL, Wallace GL. Randomized controlled effectiveness trial of executive function intervention for children on the autism spectrum. J Child Psychol Psychiatry. 2014 Apr;55(4):374-83. doi: 10.1111/jcpp.12161. Epub 2013 Nov 21. PMID 24256459
- [Background] Taylor JL, Dove D, Veenstra-VanderWeele J, et al. Comparative Effictiveness Review: Interventions for Adolescents and Young Adults With Autism. 2012;(65).
- [Background] Dingfelder HE, Mandell DS. Bridging the research-to-practice gap in autism intervention: an application of diffusion of innovation theory. J Autism Dev Disord. 2011 May;41(5):597-609. doi: 10.1007/s10803-010-1081-0. PMID 20717714
- [Background] Kenworthy L, Black DO, Harrison B, della Rosa A, Wallace GL. Are executive control functions related to autism symptoms in high-functioning children? Child Neuropsychol. 2009 Sep;15(5):425-40. doi: 10.1080/09297040802646983. PMID 19173090
- [Background] Solomon M, Ozonoff SJ, Ursu S, Ravizza S, Cummings N, Ly S, Carter CS. The neural substrates of cognitive control deficits in autism spectrum disorders. Neuropsychologia. 2009 Oct;47(12):2515-26. doi: 10.1016/j.neuropsychologia.2009.04.019. Epub 2009 May 4. PMID 19410583
- [Background] Shafritz KM, Dichter GS, Baranek GT, Belger A. The neural circuitry mediating shifts in behavioral response and cognitive set in autism. Biol Psychiatry. 2008 May 15;63(10):974-80. doi: 10.1016/j.biopsych.2007.06.028. Epub 2007 Oct 4. PMID 17916328
- [Background] Vaidya CJ, Gordon EM. Phenotypic variability in resting-state functional connectivity: current status. Brain Connect. 2013;3(2):99-120. doi: 10.1089/brain.2012.0110. PMID 23294010
- [Background] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2008 Principal Investigators; Centers for Disease Control and Prevention. Prevalence of autism spectrum disorders--Autism and Developmental Disabilities Monitoring Network, 14 sites, United States, 2008. MMWR Surveill Summ. 2012 Mar 30;61(3):1-19. PMID 22456193
- [Background] Cidav Z, Lawer L, Marcus SC, Mandell DS. Age-related variation in health service use and associated expenditures among children with autism. J Autism Dev Disord. 2013 Apr;43(4):924-31. doi: 10.1007/s10803-012-1637-2. PMID 22941343
- [Background] Shattuck PT, Narendorf SC, Cooper B, Sterzing PR, Wagner M, Taylor JL. Postsecondary education and employment among youth with an autism spectrum disorder. Pediatrics. 2012 Jun;129(6):1042-9. doi: 10.1542/peds.2011-2864. Epub 2012 May 14. PMID 22585766
- [Background] Taylor JL, Henninger NA. Frequency and correlates of service access among youth with autism transitioning to adulthood. J Autism Dev Disord. 2015 Jan;45(1):179-91. doi: 10.1007/s10803-014-2203-x. PMID 25081594
- [Background] Taylor JL, Henninger NA, Mailick MR. Longitudinal patterns of employment and postsecondary education for adults with autism and average-range IQ. Autism. 2015 Oct;19(7):785-93. doi: 10.1177/1362361315585643. Epub 2015 May 27. PMID 26019306
- [Background] Geurts HM, Verte S, Oosterlaan J, Roeyers H, Sergeant JA. How specific are executive functioning deficits in attention deficit hyperactivity disorder and autism? J Child Psychol Psychiatry. 2004 May;45(4):836-54. doi: 10.1111/j.1469-7610.2004.00276.x. PMID 15056314
- [Background] Hughes C, Russell J, Robbins TW. Evidence for executive dysfunction in autism. Neuropsychologia. 1994 Apr;32(4):477-92. doi: 10.1016/0028-3932(94)90092-2. PMID 8047253
- [Background] Ozonoff S, Pennington BF, Rogers SJ. Executive function deficits in high-functioning autistic individuals: relationship to theory of mind. J Child Psychol Psychiatry. 1991 Nov;32(7):1081-105. doi: 10.1111/j.1469-7610.1991.tb00351.x. PMID 1787138
- [Background] Ozonoff S, Jensen J. Brief report: specific executive function profiles in three neurodevelopmental disorders. J Autism Dev Disord. 1999 Apr;29(2):171-7. doi: 10.1023/a:1023052913110. No abstract available. PMID 10382139
- [Background] Kenworthy L, Yerys BE, Anthony LG, Wallace GL. Understanding executive control in autism spectrum disorders in the lab and in the real world. Neuropsychol Rev. 2008 Dec;18(4):320-38. doi: 10.1007/s11065-008-9077-7. Epub 2008 Oct 28. PMID 18956239
- [Background] Lopata C et al. ABAS-II Ratings and Correlates of Adaptive Behavior in Children with HFASDs. J Dev Phys Disabil. 2012;24:391-402.
- [Background] Lawson RA, Papadakis AA, Higginson CI, Barnett JE, Wills MC, Strang JF, Wallace GL, Kenworthy L. Everyday executive function impairments predict comorbid psychopathology in autism spectrum and attention deficit hyperactivity disorders. Neuropsychology. 2015 May;29(3):445-53. doi: 10.1037/neu0000145. Epub 2014 Oct 13. PMID 25313979
- [Background] Lounds J, Seltzer MM, Greenberg JS, Shattuck PT. Transition and change in adolescents and young adults with autism: longitudinal effects on maternal well-being. Am J Ment Retard. 2007 Nov;112(6):401-17. doi: 10.1352/0895-8017(2007)112[401:TACIAA]2.0.CO;2. PMID 17963433
- [Background] Shattuck PT, Steinberg J, Yu J, Wei X, Cooper BP, Newman L, Roux AM. Disability Identification and Self-Efficacy among College Students on the Autism Spectrum. Autism Res Treat. 2014;2014:924182. doi: 10.1155/2014/924182. Epub 2014 Feb 23. PMID 24707401
- [Background] Weisz JR, Ugueto AM, Cheron DM, Herren J. Evidence-based youth psychotherapy in the mental health ecosystem. J Clin Child Adolesc Psychol. 2013;42(2):274-86. doi: 10.1080/15374416.2013.764824. Epub 2013 Feb 12. PMID 23402704
- [Background] Ylvisaker M, Jacobs HE, Feeney T. Positive supports for people who experience behavioral and cognitive disability after brain injury: a review. J Head Trauma Rehabil. 2003 Jan-Feb;18(1):7-32. doi: 10.1097/00001199-200301000-00005. PMID 12802235
- [Background] Oberman L, Pascual-Leone A. Changes in plasticity across the lifespan: cause of disease and target for intervention. Prog Brain Res. 2013;207:91-120. doi: 10.1016/B978-0-444-63327-9.00016-3. PMID 24309252
- [Background] Lee PS, Yerys BE, Della Rosa A, Foss-Feig J, Barnes KA, James JD, VanMeter J, Vaidya CJ, Gaillard WD, Kenworthy LE. Functional connectivity of the inferior frontal cortex changes with age in children with autism spectrum disorders: a fcMRI study of response inhibition. Cereb Cortex. 2009 Aug;19(8):1787-94. doi: 10.1093/cercor/bhn209. Epub 2008 Dec 9. PMID 19068486
- [Background] Huttenlocher PR. Morphometric study of human cerebral cortex development. Neuropsychologia. 1990;28(6):517-27. doi: 10.1016/0028-3932(90)90031-i. PMID 2203993
- [Background] Giedd JN, Blumenthal J, Jeffries NO, Castellanos FX, Liu H, Zijdenbos A, Paus T, Evans AC, Rapoport JL. Brain development during childhood and adolescence: a longitudinal MRI study. Nat Neurosci. 1999 Oct;2(10):861-3. doi: 10.1038/13158. No abstract available. PMID 10491603
- [Background] Gogtay N, Giedd JN, Lusk L, Hayashi KM, Greenstein D, Vaituzis AC, Nugent TF 3rd, Herman DH, Clasen LS, Toga AW, Rapoport JL, Thompson PM. Dynamic mapping of human cortical development during childhood through early adulthood. Proc Natl Acad Sci U S A. 2004 May 25;101(21):8174-9. doi: 10.1073/pnas.0402680101. Epub 2004 May 17. PMID 15148381
- [Background] Shonkoff JP. Protecting brains, not simply stimulating minds. Science. 2011 Aug 19;333(6045):982-3. doi: 10.1126/science.1206014. PMID 21852492
- [Background] Yerys BE, Antezana L, Weinblatt R, Jankowski KF, Strang J, Vaidya CJ, Schultz RT, Gaillard WD, Kenworthy L. Neural Correlates of Set-Shifting in Children With Autism. Autism Res. 2015 Aug;8(4):386-97. doi: 10.1002/aur.1454. Epub 2015 Jan 20. PMID 25599972
- [Background] Castellanos FX, Margulies DS, Kelly C, Uddin LQ, Ghaffari M, Kirsch A, Shaw D, Shehzad Z, Di Martino A, Biswal B, Sonuga-Barke EJ, Rotrosen J, Adler LA, Milham MP. Cingulate-precuneus interactions: a new locus of dysfunction in adult attention-deficit/hyperactivity disorder. Biol Psychiatry. 2008 Feb 1;63(3):332-7. doi: 10.1016/j.biopsych.2007.06.025. Epub 2007 Sep 21. PMID 17888409
- [Background] Assaf M, Jagannathan K, Calhoun VD, Miller L, Stevens MC, Sahl R, O'Boyle JG, Schultz RT, Pearlson GD. Abnormal functional connectivity of default mode sub-networks in autism spectrum disorder patients. Neuroimage. 2010 Oct 15;53(1):247-56. doi: 10.1016/j.neuroimage.2010.05.067. Epub 2010 Jun 2. PMID 20621638
- [Background] Doyle-Thomas KA, Lee W, Foster NE, Tryfon A, Ouimet T, Hyde KL, Evans AC, Lewis J, Zwaigenbaum L, Anagnostou E; NeuroDevNet ASD Imaging Group. Atypical functional brain connectivity during rest in autism spectrum disorders. Ann Neurol. 2015 May;77(5):866-76. doi: 10.1002/ana.24391. Epub 2015 Mar 27. PMID 25707715
- [Background] Eilam-Stock T, Xu P, Cao M, Gu X, Van Dam NT, Anagnostou E, Kolevzon A, Soorya L, Park Y, Siller M, He Y, Hof PR, Fan J. Abnormal autonomic and associated brain activities during rest in autism spectrum disorder. Brain. 2014 Jan;137(Pt 1):153-71. doi: 10.1093/brain/awt294. PMID 24424916
- [Background] Jung M, Kosaka H, Saito DN, Ishitobi M, Morita T, Inohara K, Asano M, Arai S, Munesue T, Tomoda A, Wada Y, Sadato N, Okazawa H, Iidaka T. Default mode network in young male adults with autism spectrum disorder: relationship with autism spectrum traits. Mol Autism. 2014 Jun 11;5:35. doi: 10.1186/2040-2392-5-35. eCollection 2014. PMID 24955232
- [Background] Monk CS, Peltier SJ, Wiggins JL, Weng SJ, Carrasco M, Risi S, Lord C. Abnormalities of intrinsic functional connectivity in autism spectrum disorders. Neuroimage. 2009 Aug 15;47(2):764-72. doi: 10.1016/j.neuroimage.2009.04.069. Epub 2009 May 3. PMID 19409498
- [Background] Yerys BE, Gordon EM, Abrams DN, Satterthwaite TD, Weinblatt R, Jankowski KF, Strang J, Kenworthy L, Gaillard WD, Vaidya CJ. Default mode network segregation and social deficits in autism spectrum disorder: Evidence from non-medicated children. Neuroimage Clin. 2015 Aug 18;9:223-32. doi: 10.1016/j.nicl.2015.07.018. eCollection 2015. PMID 26484047
- [Background] Kennedy DP, Redcay E, Courchesne E. Failing to deactivate: resting functional abnormalities in autism. Proc Natl Acad Sci U S A. 2006 May 23;103(21):8275-80. doi: 10.1073/pnas.0600674103. Epub 2006 May 15. PMID 16702548
- [Background] Dawson G, Jones EJ, Merkle K, Venema K, Lowy R, Faja S, Kamara D, Murias M, Greenson J, Winter J, Smith M, Rogers SJ, Webb SJ. Early behavioral intervention is associated with normalized brain activity in young children with autism. J Am Acad Child Adolesc Psychiatry. 2012 Nov;51(11):1150-9. doi: 10.1016/j.jaac.2012.08.018. PMID 23101741
- [Background] Gordon I, Vander Wyk BC, Bennett RH, Cordeaux C, Lucas MV, Eilbott JA, Zagoory-Sharon O, Leckman JF, Feldman R, Pelphrey KA. Oxytocin enhances brain function in children with autism. Proc Natl Acad Sci U S A. 2013 Dec 24;110(52):20953-8. doi: 10.1073/pnas.1312857110. Epub 2013 Dec 2. PMID 24297883
- [Background] Voos AC, Pelphrey KA, Tirrell J, Bolling DZ, Vander Wyk B, Kaiser MD, McPartland JC, Volkmar FR, Ventola P. Neural mechanisms of improvements in social motivation after pivotal response treatment: two case studies. J Autism Dev Disord. 2013 Jan;43(1):1-10. doi: 10.1007/s10803-012-1683-9. PMID 23104615
- [Background] Walker HM. Use of evidence-based interventions in schools: where we've been, where we are, and where we need to go. School Psych Rev. 2004;33:398-407.
- [Background] Kasari C, Lawton K. New directions in behavioral treatment of autism spectrum disorders. Curr Opin Neurol. 2010 Apr;23(2):137-43. doi: 10.1097/WCO.0b013e32833775cd. PMID 20160648
- [Background] Pugliese CE, Anthony LG, Strang JF, Dudley K, Wallace GL, Naiman DQ, Kenworthy L. Longitudinal Examination of Adaptive Behavior in Autism Spectrum Disorders: Influence of Executive Function. J Autism Dev Disord. 2016 Feb;46(2):467-77. doi: 10.1007/s10803-015-2584-5. PMID 26349921
- [Background] J J, HA L, CK W. Subjective culture and social behavior. In: Adamopoulos J, Kashima Y, eds. Social Psychology and Cultural Context. Thousand Oaks, CA: Sage Publications; 1999:95-106.
- [Background] Wallace GL, Silvers JA, Martin A, Kenworthy LE. Brief report: Further evidence for inner speech deficits in autism spectrum disorders. J Autism Dev Disord. 2009 Dec;39(12):1735-9. doi: 10.1007/s10803-009-0802-8. Epub 2009 Jun 30. PMID 19565331
- [Background] Wechsler D, Zhou X. Wechsler Abbreviated Scale of Intelligence II. NY, New York: The Psychological Corporation: Harcourt Brace & Company; 2011.
- [Background] Lord C, Rutter M, DiLavore PC, Risi S, Gotham K, Bishop SL. Autism Diagnostic Observation Schedule, 2nd Ed. (ADOS-2). Torrance, CA: Western Psychological Services; 2012.
- [Background] Rutter M, Bailey A, Berument SK, Le Couteur A, Lord C. Social Communication Questionnaire (SCQ) Manual. Los Angeles, CA: Western Psychological Services; 2003.
- [Background] Gioia G, Isquith P, Guy S, Kenworthy L. BRIEF: Behavior Rating Inventory of Executive Function. Odessa: Psychological Assessment Resources; 2000.
- [Background] Sparrow S, Cicchetti D, Balla DA. Vineland Adaptive Behavior Scales Second Edition:Survey Forms Manual. Minneapolis, MN: Pearson; 2005.
- [Background] Abraha I, Montedori A. Modified intention to treat reporting in randomised controlled trials: systematic review. BMJ. 2010 Jun 14;340:c2697. doi: 10.1136/bmj.c2697. PMID 20547685
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Clopper CJ, Pearson ES. The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Biometrika. 1934;26:404-413.
- [Background] MATLAB Version 7.10.0. Natick, Massachusettes: The MathWorks Inc.; 2010.
- [Background] IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corporation; 2013.
- [Background] Bullmore E, Sporns O. Complex brain networks: graph theoretical analysis of structural and functional systems. Nat Rev Neurosci. 2009 Mar;10(3):186-98. doi: 10.1038/nrn2575. Epub 2009 Feb 4. PMID 19190637
- [Background] Rubinov M, Sporns O. Complex network measures of brain connectivity: uses and interpretations. Neuroimage. 2010 Sep;52(3):1059-69. doi: 10.1016/j.neuroimage.2009.10.003. Epub 2009 Oct 9. PMID 19819337
- [Background] Power JD, Cohen AL, Nelson SM, Wig GS, Barnes KA, Church JA, Vogel AC, Laumann TO, Miezin FM, Schlaggar BL, Petersen SE. Functional network organization of the human brain. Neuron. 2011 Nov 17;72(4):665-78. doi: 10.1016/j.neuron.2011.09.006. PMID 22099467
- [Background] Benjamini Y, Hochberg Y. Controlling the False Discovery Rate: A Practical and Powerful Approach to Multiple Testing. J R Stat Soc. 1995;57(1):289-300.